CLINICAL TRIAL: NCT05237479
Title: A Randomized Controlled Study Evaluating Suprainguinal Fascia Iliaca Compartment Block in Direct Anterior Approach to Total Hip Arthroplasty - A Pilot Study
Brief Title: Suprainguinal Fascia Iliaca Compartment Block in Direct Anterior Approach to Total Hip Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never approved by IRB or initiated
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-13705
Record Dates: First submitted 2022-01-10; First posted 2022-02-14 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Anesthesia, Local; Block
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: On the day of surgery, a sealed envelope with group allocation (Group A- Control vs. Group B - Intervention) will be opened by a team member not involved with data collection.
  A separate anesthesia team consisting of an anesthesiologist and certified nurse anesthetist will be responsible for the spinal anesthetic and monitored anesthesia care for both groups in the operating room A separate acute pain service team will follow the patients in both groups on postoperative day 1 and evaluate sensory and motor distribution of LFCN, FN, and ON for both groups A research assistant blinded to the allocation of both groups will collect data from the EMR for analysis. In addition, a research assistant blinded to the allocation of both groups will call patients via telephone 24 hours post-discharge for a patient satisfaction survey.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Placebo Comparator): DAA THA under spinal anesthesia ( standard of care at Montefiore)
  Interventions: Other: Placebo
- Intervention Group (Active Comparator): DAA THA under spinal anesthesia and a preoperative supra-inguinal fascia iliac compartment block (S-FICB)
  Interventions: Procedure: Suprainguinal fascia ilica block

INTERVENTIONS:
Procedure: Suprainguinal fascia ilica block — Patients who have been randomized to Group B Intervention will receive a preoperative S-FICB using 35ml of 0.5% ropivacaine under ultrasound guidance by the regional anesthesia block team once patient has been marked by surgeon. Sensory & motor distribution of the LFCN, FN, & ON will be assessed by the regional anesthesia team in the preop area for patients randomized to the control group prior to surgery. Patients who received a S-FICB in preop, approximately 15 minutes after the block, sensory & motor distribution of LFCN, FN, & ON will be assessed by the regional anesthesia block team prior to going to the operating room. All patients, regardless of group allocation, will be followed by the acute pain service team on postoperative day one to assess sensory & motor distribution of LFCN, FN, & ON & adjustment of pain medication regimens. All patients will receive a call from a research assistant blinded to group allocation 24 hours post-discharge for a patient satisfaction survey.
  Arms: Intervention Group
Other: Placebo — The sensory and motor distribution of the LFCN, FN, and ON will be assessed by the regional anesthesia team in the preop area for patients randomized to the control group prior to surgery.
  Arms: Control Group

SUMMARY:
The goal of this study is to determine whether or not a suprainguinal fascia iliaca compartment nerve block is effective at improving postoperative pain control in patients receiving an anterior approach hip replacement surgery. In general, postoperative pain control has a significant impact on earlier ambulation, initiation of physical therapy, better functional recovery, and overall patient satisfaction. The hypothesis is that providing patients with this nerve block will decrease opioid requirements in patients undergoing this surgery as compared to patients that do not receive the block.

DETAILED DESCRIPTION:
Study Design: Interventional Trial

Allocation: Randomized

Intervention Model: Parallel Assignment

Treatment groups: Group A: Control Group - DAA THA under spinal anesthesia ( standard of care at Montefiore)

Group B: Intervention Group - DAA THA under spinal anesthesia and a preoperative supra-inguinal fascia iliac compartment block (S-FICB)

Blinding Procedures:

* On the day of surgery, a sealed envelope with group allocation (Group A- Control vs. Group B - Intervention) will be opened by a team member not involved with data collection.
* For patients allocated to Group B - Intervention: A regional anesthesia block team consisting of a regional anesthesiologist, regional fellow, and resident will carry out the S-FICB in the preoperative area prior to surgery
* A separate anesthesia team consisting of an anesthesiologist and certified nurse anesthetist will be responsible for the spinal anesthetic and monitored anesthesia care for both groups in the operating room
* A separate acute pain service team will follow the patients in both groups on postoperative day 1 and evaluate sensory and motor distribution of LFCN, FN, and ON for both groups
* A research assistant blinded to the allocation of both groups will collect data from the EMR for analysis. In addition, a research assistant blinded to the allocation of both groups will call patients via telephone 24 hours post-discharge for a patient satisfaction survey.

Hypothesis: The supra-inguinal fascia iliaca compartment block will decrease 24 hours post-surgery opioid requirements in patients undergoing elective direct anterior approach to total hip arthroplasty.

Target Population: Patients undergoing primary elective total hip arthroplasty under direct anterior surgical approach

Recruitment methods: Participants who meet the inclusion/exclusion criteria for the study will be approached to participate in the study at the preoperative visit at the Orthopedic Surgeon's Office. Informed consent for participation in the study will be obtained during the preoperative visit.

The planned interventions and their timing:

* On the day of surgery, patients who have been randomized to Group B - Intervention will receive a preoperative S-FICB using 35 ml of 0.5% ropivacaine (max dose of 3mg/kg) under ultrasound guidance by the regional anesthesia block team once the patient has been marked by the surgeon
* The sensory and motor distribution of the LFCN, FN, and ON will be assessed by the regional anesthesia team in the preop area for patients randomized to the control group prior to surgery. For those patients who received a S-FICB in preop, approximately 15 minutes after the block, sensory and motor distribution of LFCN, FN, and ON will be assessed by the regional anesthesia block team prior to going to the operating room.
* All patients, regardless of group allocation, will be followed by the acute pain service team on postoperative day one to assess sensory and motor distribution of LFCN, FN, and ON and adjustment of pain medication regimens
* All patients will receive a telephone call from a research assistant blinded to group allocation 24 hours post-discharge for a patient satisfaction survey.
* Postoperatively all patients will be placed on the following pain regimen:
* All patients will be started on a Hydromorphone intravenous patient-controlled analgesia (PCA) for 24 hours, with starting parameters: 0.2mg q10 min bolus dosing without a basal rate.
* A standardized regimen of non-opioid adjuvants will include: Acetaminophen 975mg po q8h, Pregabalin 50mg po BID, Ketorolac 15mg q8h IV x 24 hours followed by Celebrex 200mg po BID.
* After the first 24 hours, patients will be transitioned off the hydromorphone PCA with oxycodone 5mg PO q4h prn for moderate pain and 10mg PO q4h prn for severe pain, hydromorphone 0.2mg IV q4h prn for breakthrough pain. These doses may be increased or decreased thereafter at the discretion of the acute pain service team based on patient evaluation and reported pain scores.

Study Population

A. Patients undergoing elective primary total hip arthroplasty under direct anterior surgical approach with neuraxial anesthesia

Participant Recruitment

Participants will be recruited during their preoperative visit to the office of the orthopedic surgery team performing the patient's surgery. At this visit, where the patient will be consented for the surgery itself, the orthopedic surgery team will present the opportunity to participate in this study during the perioperative period to patients who meet inclusion/exclusion criteria. The informed consent document will be presented to the patient at this time for review. Contact information to the study's primary investigator and anesthesia associates will be provided on the informed consent documentation if the patient should require any further information about the study. If after reviewing the study details in the consent documentation, the patient is amenable to participating, they may provide consent by signing the consent form at the orthopedic surgeon's office free from coercion. Following enrollment in the study, patient data will be collected by the primary investigator's research team, stored securely, and all patient information and data will be de-identified prior to publication.

Risks/Benefits Anticipated risks of this study include the risks associated with the S-FICB procedure itself. These include infection, bleeding, injury to surrounding structures including nerves, and local anesthetic systemic toxicity which can occur if a large amount of local anesthetic is inadvertently injected intravascularly. This procedure is performed under sterile conditions, minimizing the risk of infection. In addition, patients who have local infection at the site of injection will be excluded as participants. The risks of major bleeding is rare for patients who do not have preexisting coagulopathies, and is low for patients who are on anticoagulation that has been discontinued an appropriate amount of time prior to surgery according to the American Society for Regional Anesthesia (ASRA) guidelines. Furthermore, the risk of nerve injury is greatly mitigated using ultrasound guidance in performing this type of nerve block where nerve tissue can be identified visually. Additionally, because this is a fascial plane block, the investigators do not aim to inject local anesthetic directly adjacent to nerve structures, minimizing risk of nerve injury or damage. The use of ultrasound guidance also mitigates the risk of local anesthetic systemic toxicity as blood vessels can be visualized and avoided. The practice of frequent aspiration during injection of local anesthetic also protects against this risk.

Another risk to participants of this study is the possible loss of confidentiality; however, the investigators have designed this study to include protocols for keeping patient information private. In addition, strict storage and de-identification of data will be used to protect patient information.

This study presents several possible benefits to participants and future patients who must undergo this surgery. It presents a potential avenue for decreasing opioid requirements in the perioperative period. Adverse events associated with opioids cause significant morbidity to the patient in the postoperative period. These include nausea, vomiting, sedation and dizziness that can lead to falls during attempted ambulation and inability to participate in physical therapy, and respiratory depression requiring intervention. All of these possible events can hinder recovery significantly and contribute to longer hospital lengths of stay.

Improved pain control overall is also a potential benefit to patients participating in this study. Decreasing the levels of pain experienced by patients is often instrumental in improving a patient's satisfaction with their surgery and in-hospital recovery. Decreased pain also makes it less challenging for a patient to participate fully in physical therapy, aiding in the recovery process after major orthopedic surgery.

If the results of this study support the use of the S-FICB showing improved outcomes for patients in the postoperative period, this peripheral nerve block can be more widely employed and incorporated as part of a multimodal perioperative opioid sparing pathway to improve outcomes for this patient population in the future.

The S-FICB is a relatively low-risk procedure, while the potential benefits to participants in this study, as well as future participants, is substantial.

Randomization On the day of surgery, an envelope containing the randomization code will be given to the regional team responsible for the study patient. Patients will be randomly allocated to receive S-FICB or standard of care using a 1:1 allocation ratio. --- BMI.--- A research associate who is not directly involved with the study procedures will maintain the randomization codes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary elective total hip arthroplasty under direct anterior surgical approach
* ASA Class I-III
* Age > 18 years old

Exclusion Criteria:

Patient refusal

* Inability to understand and sign an informed consent
* Infection at the injection site
* Allergy or hypersensitivity to ropivacaine or other amide local anesthetics
* Contraindication or patient refusal to get spinal anesthesia
* Thrombocytopenia (Platelets < 100, 000)
* Coagulopathy (INR > 1.4)
* Use of anticoagulant drugs that have not been discontinued in an appropriate amount of time - according to American Society of Regional Anesthesia guidelines, prior to surgery
* End-Stage Renal Disease
* ASA Class IV-V
* Patients on chronic opioid therapy on most days for > 3 months [19].
* BMI>40

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphine Milligram Equivalent (MME) | In PACU (1-2 hours postoperatively)
  Morphine Milligram Equivalent use in PACU
Morphine Milligram Equivalent (MME) | 24 hours postoperatively
  Morphine Milligram Equivalent use post-op

SECONDARY OUTCOMES:
Sensory and Motor Distribution of LFCN, FN and ON | Preoperatively prior to surgery
  Sensory assessment of the LCFN, FN and ON - Response to pinprick in the anterior, medial and lateral aspects of the thigh Motor assessment of FN and ON - To test FN: Investigator supports knee under popliteal fossa and patient is asked to extend knee against resistance.
  To test ON: Patient's leg is abducted in the supine position and patient will be asked to adduct knee to the midline.
  Sensory assessment of the LCFN, FN and ON - Response to pinprick in the anterior, medial and lateral aspects of the thigh Motor assessment of FN and ON - To test FN: Investigator supports knee under popliteal fossa and patient is asked to extend knee against resistance.
  To test ON: Patient's leg is abducted in the supine position and patient will be asked to adduct knee to the midline.
Sensory and Motor Distribution of LFCN, FN and ON | Postoperatively 24 hours after surgery
  Sensory assessment of the LCFN, FN and ON - Response to pinprick in the anterior, medial and lateral aspects of the thigh Motor assessment of FN and ON - To test FN: Investigator supports knee under popliteal fossa and patient is asked to extend knee against resistance.
  To test ON: Patient's leg is abducted in the supine position and patient will be asked to adduct knee to the midline.
  Sensory assessment of the LCFN, FN and ON - Response to pinprick in the anterior, medial and lateral aspects of the thigh Motor assessment of FN and ON - To test FN: Investigator supports knee under popliteal fossa and patient is asked to extend knee against resistance.
  To test ON: Patient's leg is abducted in the supine position and patient will be asked to adduct knee to the midline.
Length of Hospital Stay | Up to 7 days
  To determine the average length of hospital stay (LOS) in Group A - control (did not receive the S-FICB) and Group B: Intervention (received S-FICB)
Patient satisfaction of acute postoperative pain management experience | 24 hours post discharge
  Ordinal variables consisting of varying levels of satisfaction namely: Very satisfied, Satisfied, Somewhat Satisfied, Unsatisfied, and Very Unsatisfied
Pain scores in PACU | PACU stay
  Numerical Pain rating, scale of 0-10
Pain scores at 24 hours Postoperatively | 24 hours postoperatively
  Numerical Pain rating, scale of 0-10
Pain scores at 48 hours Postoperatively | 48 hours
  Numerical Pain rating, scale of 0-10
Emergency Department Readmissions postoperatively | 1-7 days postoperatively
  Emergency department visit or readmission within 7 days following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia steinberg, DO, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kloppenburg M, Berenbaum F. Osteoarthritis year in review 2019: epidemiology and therapy. Osteoarthritis Cartilage. 2020 Mar;28(3):242-248. doi: 10.1016/j.joca.2020.01.002. Epub 2020 Jan 13. PMID 31945457
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Zhang D, Pan L, Maimaitijuma T, Liu H, Wu H. Imaging Analysis of Prosthesis Angle after Hip Replacement with Direct Anterior Approach in Lateral Position. J Healthc Eng. 2021 Feb 17;2021:5540834. doi: 10.1155/2021/5540834. eCollection 2021. PMID 33680413
- [Background] Galakatos GR. Direct Anterior Total Hip Arthroplasty. Mo Med. 2018 Nov-Dec;115(6):537-541. PMID 30643349
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Kumar K, Kirksey MA, Duong S, Wu CL. A Review of Opioid-Sparing Modalities in Perioperative Pain Management: Methods to Decrease Opioid Use Postoperatively. Anesth Analg. 2017 Nov;125(5):1749-1760. doi: 10.1213/ANE.0000000000002497. PMID 29049119
- [Background] Bugada D, Bellini V, Lorini LF, Mariano ER. Update on Selective Regional Analgesia for Hip Surgery Patients. Anesthesiol Clin. 2018 Sep;36(3):403-415. doi: 10.1016/j.anclin.2018.04.001. Epub 2018 Jul 11. PMID 30092937
- [Background] Xia Q, Ding W, Lin C, Xia J, Xu Y, Jia M. Postoperative pain treatment with transmuscular quadratus lumborum block and fascia iliaca compartment block in patients undergoing total hip arthroplasty: a randomized controlled trial. BMC Anesthesiol. 2021 Jul 10;21(1):188. doi: 10.1186/s12871-021-01413-7. PMID 34243719
- [Background] Nassar H, Hasanin A, Sewilam M, Ahmed H, Abo-Elsoud M, Taalab O, Rady A, Zoheir HA. Transmuscular Quadratus Lumborum Block versus Suprainguinal Fascia Iliaca Block for Hip Arthroplasty: A Randomized, Controlled Pilot Study. Local Reg Anesth. 2021 Apr 20;14:67-74. doi: 10.2147/LRA.S308964. eCollection 2021. PMID 33907462
- [Background] Desmet M, Balocco AL, Van Belleghem V. Fascia iliaca compartment blocks: Different techniques and review of the literature. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):57-66. doi: 10.1016/j.bpa.2019.03.004. Epub 2019 Apr 17. PMID 31272654
- [Background] O'Reilly N, Desmet M, Kearns R. Fascia iliaca compartment block. BJA Educ. 2019 Jun;19(6):191-197. doi: 10.1016/j.bjae.2019.03.001. Epub 2019 Apr 24. No abstract available. PMID 33456890
- [Background] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Background] Dolan J, Williams A, Murney E, Smith M, Kenny GN. Ultrasound guided fascia iliaca block: a comparison with the loss of resistance technique. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):526-31. doi: 10.1016/j.rapm.2008.03.008. PMID 19258967
- [Background] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Background] Vermeylen K, Desmet M, Leunen I, Soetens F, Neyrinck A, Carens D, Caerts B, Seynaeve P, Hadzic A, Van de Velde M. Supra-inguinal injection for fascia iliaca compartment block results in more consistent spread towards the lumbar plexus than an infra-inguinal injection: a volunteer study. Reg Anesth Pain Med. 2019 Feb 22:rapm-2018-100092. doi: 10.1136/rapm-2018-100092. Online ahead of print. PMID 30798268
- [Background] Zhang XY, Ma JB. The efficacy of fascia iliaca compartment block for pain control after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Jan 25;14(1):33. doi: 10.1186/s13018-018-1053-1. PMID 30683117
- [Background] Desmet M, Vermeylen K, Van Herreweghe I, Carlier L, Soetens F, Lambrecht S, Croes K, Pottel H, Van de Velde M. A Longitudinal Supra-Inguinal Fascia Iliaca Compartment Block Reduces Morphine Consumption After Total Hip Arthroplasty. Reg Anesth Pain Med. 2017 May/Jun;42(3):327-333. doi: 10.1097/AAP.0000000000000543. PMID 28059869
- [Background] Flevas DA, Tsantes AG, Mavrogenis AF. Direct Anterior Approach Total Hip Arthroplasty Revisited. JBJS Rev. 2020 Apr;8(4):e0144. doi: 10.2106/JBJS.RVW.19.00144. PMID 32304500
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Background] Memtsoudis SG, Poeran J, Cozowicz C, Zubizarreta N, Ozbek U, Mazumdar M. The impact of peripheral nerve blocks on perioperative outcome in hip and knee arthroplasty-a population-based study. Pain. 2016 Oct;157(10):2341-2349. doi: 10.1097/j.pain.0000000000000654. PMID 27643835